CLINICAL TRIAL: NCT05006560
Title: An Internet-based Rehabilitation Aftercare Program Focusing on Physical Activity Promotion for Persons With Chronic Obstructive Pulmonary Disease
Brief Title: Internet-based Rehabilitation Aftercare Focusing on Physical Activity Promotion in Persons With COPD
Acronym: COPD-AReNa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Bad Reichenhall Clinic, Center for Rehabilitation, Pulmonology and Orthopedics German Statutory Pension Insurance (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Head of the Department of Sport Science and Sport, University of Erlangen-Nürnberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F010-2020
Record Dates: First submitted 2021-07-31; First posted 2021-08-16 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; exercise; physical activity promotion; behavior change; internet-based intervention; physical literacy; rehabilitation aftercare; mhealth; telerehabilitation; feasibility
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care rehabilitation and aftercare (Experimental): Participants receive the standard inpatient pulmonary rehabilitation followed by an internet based 12-week rehabilitation aftercare program.
  Interventions: Other: Pulmonary Rehabilitation (usual care); Other: After care: Exercise and physical activity promotion
- Rehabilitation and aftercare (aligned) (Experimental): Participants receive the standard inpatient pulmonary rehabilitation followed by an internet based 12-week rehabilitation aftercare program.
  During rehabilitation, participants already get familiarized with components of the after care program.
  Interventions: Other: Pulmonary Rehabilitation (usual care) + familiarization with components of the aftercare program; Other: After care: Exercise and physical activity promotion

INTERVENTIONS:
Other: Pulmonary Rehabilitation (usual care) — Participants receive the standard inpatient pulmonary rehabilitation (PR) in a specialized German Rehabilitation Clinic. PR is a comprehensive, multidisciplinary intervention implemented by an interdisciplinary rehabilitation team. PR is based on a patient assessment followed by a combination of patient-tailored therapies. PR includes the following obligatory main components: Checking and, if required, adjusting the current COPD medication according to current guidelines; physical training (endurance training, strength training, whole body vibration muscle training); structured education; respiratory physiotherapy. PR lasts on average 25 days.
  Arms: Usual care rehabilitation and aftercare
Other: Pulmonary Rehabilitation (usual care) + familiarization with components of the aftercare program — Participants receive the standard inpatient pulmonary rehabilitation (PR) in a specialized German Rehabilitation Clinic. PR is a comprehensive, multidisciplinary intervention implemented by an interdisciplinary rehabilitation team. PR is based on a patient assessment followed by a combination of patient-tailored therapies. PR includes the following obligatory main components: Checking and, if required, adjusting the current COPD medication according to current guidelines; physical training (endurance training, strength training, whole body vibration muscle training); structured education; respiratory physiotherapy. PR lasts on average 25 days. Additionally, participants use several functions of the aftercare program's mobile application. This includes using the application during endurance and strength training (as part of usual care) and using a consumer activity monitor to count daily steps.
  Arms: Rehabilitation and aftercare (aligned)
Other: After care: Exercise and physical activity promotion — Participants will agree with their therapist on an exercise plan (endurance and resistance training) that are made available for participants through the study's mobile app. Frequency and duration of endurance and strength training are prescribed in accordance with exercise guidelines for persons with COPD. However, they can be adjusted according to participants needs.
  Next to the exercise, participants receive physical activity counseling. This consists of phone or video calls with a therapist, group video calls with a therapist, a complementary e-learning course as well as complementary functions of the study's mobile app.

SUMMARY:
The aim of the study is to evaluate a 12-week internet-based rehabilitation aftercare program with an emphasis on physical activity promotion for persons with COPD. The program starts directly after an inpatient pulmonary rehabilitation program. It includes monitoring and promotion of physical activity, progressive resistance and endurance training, education through online learning modules and continuous support from a therapist.

ELIGIBILITY:
Inclusion Criteria:

* Main diagnosis for the Pulmonary Rehabilitation is an International Classification of Diseases-Code J44.- (Other chronic obstructive pulmonary disease) at all 2011 Global Initiative for Chronic Obstructive Lung Disease (GOLD) classifications A-D and stages 1-4.
* Internet access at home
* owning a smartphone with the operating system Android or iOS
* basic computer and internet skills (e. g. using web browser)
* ability to operate a smartphone (especially to install mobile applications)
* ability to read, write and comprehend as well as communicate electronically

Exclusion Criteria:

* severe concomitant disease, which will affect the ability to be physically active more than COPD for example, cancer or severe cardiac, neurological, orthopaedic or metabolic comorbidities)
* cognitive impairment that hampers study implementation
* Lack of ability to speak German

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the intervention and participants' satisfaction (participant perspective) | one week after the rehabilitation aftercare program (T2)
  Semi-structured interviews will be conducted with persons with COPD that participated in the study.
Acceptability and practicability of intervention (therapist perspective) | one week after the last participant was supervised by the therapist
  Semi-structured interviews will be conducted with therapists that delivered the intervention.
Recruitment | 6 to 3 weeks prior to inpatient rehabilitation
  Number of participants screened, number of eligible participants, number of participants recruited, reasons for exclusion during recruitment
Compliance with intervention protocol | from the start of the aftercare program, until the end of the aftercare program, on average 12 weeks
  Completed training sessions, e-learning modules and telephone calls with the therapist will be documented for each participant.
Retention | one week after the rehabilitation aftercare program (T2)
  Percentage of included participants that complete T2 assessment.

SECONDARY OUTCOMES:
Dyspnea, cough, sputum, pain | Two weeks prior to inpatient rehabilitation (T-1), during the last week of pulmonary rehabilitation (T1), one week after the rehabilitation aftercare program (T2)
  Questionnaire: Numeric Rating Scales (self-developed)
  The questionnaire consists of seven items. Items can be answered on a eleven-step numeric rating scale (0-10). Items are analyzed individually.
COPD Assessment Test (CAT) | Two weeks prior to inpatient rehabilitation (T-1), during the last week of pulmonary rehabilitation (T1), one week after the rehabilitation aftercare program (T2)
  Questionnaire: Impact of COPD on health status
  The questionnaire consists of eight questions that can be answered on a six-point likert scale (0-5). All answers are added up to determine the overall score (0 to 40). Higher scores indicate that COPD has more impact on the participant's life.
St. Georges Respiratory Questionnaire (SGRQ) (4 weeks) | Two weeks prior to inpatient rehabilitation (T-1), during the last week of pulmonary rehabilitation (T1), one week after the rehabilitation aftercare program (T2)
  Questionnaire: Overall health, daily life, and perceived well-being in patients with obstructive airways disease
  The questionnaire consists of 52 items. The overall score ranges from 0-100, with higher scores indicating more limitations.
Patient Health Questionnaire (PHQ-9) | Two weeks prior to inpatient rehabilitation (T-1), during the last week of pulmonary rehabilitation (T1), one week after the rehabilitation aftercare program (T2)
  Questionnaire: Depression
  The questionnaire consists of 9 items that can be answered on a 4-point likert scale (0-3 points). Answers are added to a sum score, with higher scores indicating higher depression levels.
COPD-Anxiety Questionnaire (CAF-R) | Two weeks prior to inpatient rehabilitation (T-1), during the last week of pulmonary rehabilitation (T1), one week after the rehabilitation aftercare program (T2)
  Questionnaire: COPD specific fears
  The CAF-R consists of 20-items that are rated on a 5-point Likert-type scale (0= never to 4=always). Five scales can be built: fear of dyspnea, fear of physical activity, fear of progression, fear of social exclusion, and sleep-related worries. Additionally, an overall score can be calculated (sum of all items).
Physical activity-related health competence questionnaire | During the first week of pulmonary rehabilitation (T0), during the last week of pulmonary rehabilitation (T1), one week after the rehabilitation aftercare program (T2)
  42-item questionnaire that measures physical activity-related health competence. The physical activity related health competence consists of three subcompetencies: movement competence (18 items), control competence (10 items), physical activity-related self-regulation competence (14 items). Scores for each subcompetence can be calculated as sum scores, mean scores, or percentages. Higher scores indicate higher levels of the subcompetences.
BSA-Questionnaire | Two weeks prior to inpatient rehabilitation (T-1), during the last week of pulmonary rehabilitation (T1), one week after the rehabilitation aftercare program (T2)
  Questionnaire: Subjectively measured physical activity
  The questionnaire asks for physical activities during a typical week. It differentiates between leisure-time/transportation activities (physical activity score) and sport-/exercise-related activities (sports score). Participants are required to report frequency and duration of activities executed during the last two weeks. Minutes of leisure-time physical activity per week and sport-/exercise related activity per week are calculated to get the physical activity and the sports score. Both scores can be combined in order to receive the overall volume of physical activity completed during leisure-time and transportation as well as sport-/exercise-related activities.
Bief Fatigue Inventory (BFI) | Two weeks prior to inpatient rehabilitation (T-1), during the last week of pulmonary rehabilitation (T1), one week after the rehabilitation aftercare program (T2)
  Questionnaire: Fatigue
  The BFI starts with a question asking the patient whether he feels more than usual fatigued or tired (yes/no). This question is followed by nine items on the intensity of fatigue as well as impairments caused by fatigue. These questions can be answered on an eleven-step numerical rating scale (0-10), with higher scores indicating higher intensity and impairment. The total BFI score is the mean of the nine items.
Health Care Climate Questionnaire (German version) (HCCQ-D) | during the last week of pulmonary rehabilitation (T1), one week after the rehabilitation aftercare program (T2)
  Questionnaire: patients' perceived autonomy support from their health care provider
  The questionnaire consists of 15 items that can be answered on a seven-point Likert scale (1=strongly disagree, 7=strongly agree). An overall score is calculated by taking the average of individual item scores.
Usability and usefulness of the mobile application (meCue 2.0 questionnaire) | during the last week of pulmonary rehabilitation (T1) (only intervention group), one week after the rehabilitation aftercare program (T2)
  The module usability and usefulness of the meCue 2.0 questionnaire was used. The module contains 3 items on usability and 3 items on usefulness that are answered on a 7-point Likert scale (scored from 1 to 7). In order two receive a score for usability and a score for usefulness, the mean is calculated for the items of each area

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pfeifer, Prof. Dr., Principal Investigator — Friedrich-Alexander University Erlangen-Nürnberg; Konrad Schultz, Dr. med., Principal Investigator — Bad Reichenhall Clinic, Center for Rehabilitation, Pulmonology and Orthopedics German Statutory Pension Insurance
Locations (1):
- Klinik Bad Reichenhall der Deutschen Rentenversicherung Bayern Süd, Bad Reichenhall, Germany